CLINICAL TRIAL: NCT07377097
Title: Effects of Sweetener Consumption on Risk Factors for Heart Disease
Brief Title: Effects of Sweetener Consumption on Risk Factors for Heart Disease in Prediabetic Subjects
Acronym: Sweetheart
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Marco Witkowski, Marco Witkowski, MD, PhD, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: Sweetheart-Study
Record Dates: First submitted 2025-12-11; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-12

CONDITIONS: Prediabetic State; Metabolic Syndrome; Insulin Resistance; Thrombosis; Hypercoagulable State; Cardiovascular (CV) Risk; Cardiovascular Risk Factors; Cardiovascular Diseases (CVD); Prediabetes; Prediabetes / Type 2 Diabetes; Sweeteners
MeSH Terms: conditions — Prediabetic State; Metabolic Syndrome; Insulin Resistance; Thrombosis; Thrombophilia; Cardiovascular Diseases; Diabetes Mellitus, Type 2 | interventions — Saccharin; trichlorosucrose; Erythritol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Saccharin Group (Active Comparator): Intervention: Saccharin
  Interventions: Dietary Supplement: Saccharin
- Sucralose Group (Active Comparator): Intervention: Sucralose
  Interventions: Dietary Supplement: Sucralose
- Erythritol Group (Active Comparator): Intervention: Erythritol
  Interventions: Dietary Supplement: Erythritol
- Control Group (Placebo Comparator): Intervention: Vehicle
  Interventions: Dietary Supplement: Vehicle

INTERVENTIONS:
Dietary Supplement: Saccharin — Participants in the saccharin group will consume 5 mg/kg body weight of saccharin daily, dissolved in 500 mL of water. This corresponds to the maximum recommended daily intake as determined by EFSA and JECFA (the joint FAO/WHO Expert Committee on Food Additives).
  Arms: Saccharin Group
Dietary Supplement: Sucralose — Participants in the sucralose group will consume 15 mg/kg body weight of sucralose daily in 500 mL of water, representing the maximum recommended daily intake.
  Arms: Sucralose Group
Dietary Supplement: Erythritol — Those in the erythritol group will consume 0.5 g/kg body weight of erythritol daily in 500 mL of water, a dose considered safe and below levels that cause digestive discomfort (European Food Safety Authority [EFSA], 2023).
  Arms: Erythritol Group
Dietary Supplement: Vehicle — Participants in the control group (vehicle) will receive a vehicle consisting of 500 mL unsweetened lemon soda
  Arms: Control Group

SUMMARY:
The aim of this prospective interventional study is to investigate the metabolic effects of consuming artificial and natural sweeteners in persons with prediabetes. Prediabetes is a condition characterized by blood sugar levels that are elevated above normal but not yet meeting the criteria for type 2 diabetes. This condition markedly increases the risk of progressing to type 2 diabetes, which in turn can lead to complications including cardiovascular diseases.

Artificial sweeteners such as saccharin and sucralose, as well as natural sugar substitutes like erythritol, are increasingly used as alternatives to sugar and are recommended for individuals at cardiometabolic risk - including overweight individuals, patients with prediabetes, or diabetics - to help reduce caloric intake. Recent literature has reported possible negative associations between artificial sweeteners and blood sugar regulation in healthy subjects (1). Additionally, effects on various blood cells have been observed. For example, erythritol has been shown to alter platelet function leading to increased reactivity in healthy study participants following consumption (2).

However, the impact of alternative sweeteners on metabolic processes and their effects on blood coagulation in patients with prediabetes-a population at increased risk-has not been systematically studied. In this planned interventional study, 80 patients meeting laboratory criteria for prediabetes will be randomly assigned to one of four groups, each receiving a different intervention for two weeks: saccharin, sucralose, erythritol, or a control group receiving water. The doses reflect the acceptable daily intake or known doses that are considered safe.

After enrollment, participants will visit the study center 2 times: before starting the intervention and after completing the intervention. During these visits, biological samples such as blood, urine, and stool will be collected to study metabolism, gut bacteria, immune and blood cell function. Tests will include an oral glucose tolerance test, coagulation tests, and additional blood analyses. Additionally, participants will wear a glucose monitor to track blood sugar fluctuations during the intervention.

The investigators hypothesize that consumption of alternative sweeteners negatively affects blood sugar regulation and insulin sensitivity in patients with prediabetes. Furthermore, this study will explore how the candidate sweeteners influence the gut microbiome, blood cells and other metabolic factors in this population.

ELIGIBILITY:
Inclusion Criteria:

* Presence of prediabetes (HbA1c 5.7-6.4% or glucose after oral glucose tolerance test 140 to 199 mg/dL)
* Written informed consent available

Exclusion Criteria:

* Inability to communicate sufficiently in the required language
* Dementia or other significantly cognitively impairing condition
* Current pregnancy or breastfeeding
* Other severe internal, neurological, or psychiatric condition
* History of gout
* History of gallstones / diagnosis of cholelithiasis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-01-05 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Change of glucose tolerance | Baseline vs. within 1 week after intervention
  Measured by AUC of oral glucose tolerance test

SECONDARY OUTCOMES:
Change of microbiome | Baseline vs. within 1 week after intervention
  RNA-Sequencing of stool samples
Flow cytometry analysis of changes in frequency of circulating monocyte subsets (%) | Baseline vs. within 1 week after intervention
  Measured by flow cytometry in isolated PBMCs (Peripheral Blood Mononuclear Cells) using specific antibodies with binding to CD45, CD14, CD15 and CD16 to define monocyte subsets. Values will be reported as percent of CD45+ leukocytes
Flow cytometry analysis of changes in platelet activation marker expression (% positive platelets) | Baseline vs. within 1 week after intervention
  Whole blood samples will be analyzed using flow cytometry. Platelets will be detected based on size and using well-established surface markers (CD41). Activation markers will be assessed (CD62P and PAC1) and reported as percent of positive cells.
Flow cytometry analysis of changes in platelet activation marker expression (MFI) | Baseline vs. within 1 week after intervention
  Whole blood samples will be analyzed using flow cytometry. Platelets will be detected based on size and using well-established surface markers (CD41). Activation markers will be assessed (CD62P and PAC1) and reported as mean fluorescence intensity.
Changes in lipid profile | Baseline vs. within 1 week after intervention
  Serum analysis of Total cholesterol, HDL and LDL cholesterol, triglycerides
Changes in blood metabolite profiles by liquid chromatography / mass spectrometry | Baseline vs. within 1 week after intervention
  Untargeted metabolomics analysis of plasma samples using liquid chromatography-mass spectrometry (LC/MS). Data will be reported as relative ion intensity changes from baseline (log2 fold change, mean ± SD) for significantly altered features.
Changes in body mass index (BMI) | Baseline vs. within 1 week after intervention
  To observe changes in anthropometric measures. Measurement of height in meters and weight in kilograms to calculate body mass index (BMI = weight/height^2) in kg/m^2
Changes in waist to hip ratio (WHR) | Baseline vs. within 1 week after intervention
  To observe changes in anthropometric measures. Measurement of waist circumference and hip circumference to calculate waist-to-hip-ratio WHR (waist circumference divided by hip circumference).
Changes in body fat percentage | Baseline vs. within 1 week after intervention
  Measured by Bioelectrical Impedance Analysis (BIA)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Witkowski M, Wilcox J, Province V, Wang Z, Nemet I, Tang WHW, Hazen SL. Ingestion of the Non-Nutritive Sweetener Erythritol, but Not Glucose, Enhances Platelet Reactivity and Thrombosis Potential in Healthy Volunteers-Brief Report. Arterioscler Thromb Vasc Biol. 2024 Sep;44(9):2136-2141. doi: 10.1161/ATVBAHA.124.321019. Epub 2024 Aug 8. PMID 39114916
- [Background] Suez J, Cohen Y, Valdes-Mas R, Mor U, Dori-Bachash M, Federici S, Zmora N, Leshem A, Heinemann M, Linevsky R, Zur M, Ben-Zeev Brik R, Bukimer A, Eliyahu-Miller S, Metz A, Fischbein R, Sharov O, Malitsky S, Itkin M, Stettner N, Harmelin A, Shapiro H, Stein-Thoeringer CK, Segal E, Elinav E. Personalized microbiome-driven effects of non-nutritive sweeteners on human glucose tolerance. Cell. 2022 Sep 1;185(18):3307-3328.e19. doi: 10.1016/j.cell.2022.07.016. Epub 2022 Aug 19. PMID 35987213